CLINICAL TRIAL: NCT05287152
Title: Titanium Tacked Soft Tissue Stabilization : A Novel Technique For Free Gingival Graft Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Mohamed Khairy Mohammed Tammam, A dentist in oral implantology department ( master degree), Egyptian Biomedical Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: free gingival graft fixation
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Lack of Keratinized Gingiva

STUDY DESIGN:
Intervention Model Description: Using the titanium tacks in free gingival graft fixation instead of conventional suturing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: titanium tacks or pins — using tacks or pins made of titanium 2.5 mm diameter and 4mm length for free gingival graft fixation.

SUMMARY:
A case series study on ten patients with lack of keratinization in the non-esthetic area .the purpose of the study is the evaluation of using the titanium tacks in free gingival graft fixation as an alternative to the conventional suturing techniques or the tissue adhesives.

DETAILED DESCRIPTION:
A case series study conducted on 10 patients with lack of keratinization in the non- esthetic areas for clinical evaluation of the effeciancy of the titanium tacks in free gingival graft fixation in terms of the amount of the graft shrinkage through out a six months follow up period . the records will be taken through imagej software for comparing the graft surface area at 1 , 3 and six months .

ELIGIBILITY:
Inclusion Criteria:

* patient with lack of keratinization in the non-esthetic areas

Exclusion Criteria:

* patients on chemotherapy
* patients on radiotherapy
* smokers
* patients with bad oral hygiene

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
evaluation of the amount of the free gingival graft contraction when being fixed using the titanium tacks( bone tacks) | 6 months
  evaluating the amount of graft contraction by a software standardized surface area calibration of digital photographs taken at one, three, and six months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Od Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thoma DS, Naenni N, Figuero E, Hammerle CHF, Schwarz F, Jung RE, Sanz-Sanchez I. Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:32-49. doi: 10.1111/clr.13114. PMID 29498129
- [Result] Dragan IF, Hotlzman LP, Karimbux NY, Morin RA, Bassir SH. Clinical Outcomes of Comparing Soft Tissue Alternatives to Free Gingival Graft: A Systematic Review and Meta-Analysis . J Evid Based Dent Pract. 2017 Dec;17(4):370-380.e3. doi: 10.1016/j.jebdp.2017.05.008. Epub 2017 May 26. PMID 29197438
- [Result] Lim HC, An SC, Lee DW. A retrospective comparison of three modalities for vestibuloplasty in the posterior mandible: apically positioned flap only vs. free gingival graft vs. collagen matrix. Clin Oral Investig. 2018 Jun;22(5):2121-2128. doi: 10.1007/s00784-017-2320-y. Epub 2017 Dec 23. PMID 29275490
- [Result] Greenwell H, Fiorellini J, Giannobile W, Offenbacher S, Salkin L, Townsend C, Sheridan P, Genco R; Research, Science and Therapy Committee. Oral reconstructive and corrective considerations in periodontal therapy. J Periodontol. 2005 Sep;76(9):1588-600. doi: 10.1902/jop.2005.76.9.1588. PMID 16171452
- [Result] Korkis S, Thompson TN, Vizirakis MA, Lamble M, Zimmerman D, Neely AL, Kinaia BM. Stabilization Techniques for Soft Tissue Grafting Around Dental Implants: Case Report. Clin Adv Periodontics. 2019 Dec;9(4):192-195. doi: 10.1002/cap.10071. Epub 2019 Sep 23. PMID 31497932
- [Result] Shi Y, Segelnick SL, El Chaar ES. A Modified Technique of Tacking Acellular Dermal Matrix to Increase Keratinized Mucosa Around Dental Implants as an Alternative to a Free Gingival Graft: A Case Report. Clin Adv Periodontics. 2020 Dec;10(4):175-180. doi: 10.1002/cap.10113. Epub 2020 Aug 13. PMID 32692900